CLINICAL TRIAL: NCT03851276
Title: A Multicentre, Single Arm Pilot Study to Evaluate the Safety and the Feasibility of Planning and Execution of Surgical Revascularization in Patients With Complex Coronary Artery Disease, Based Solely on Non-invasive MSCT Angiography Imaging Utilizing High-definition GE Healthcare RevolutionTM CT and HeartFlow FFRCT.
Brief Title: A Multicentre, Pilot Study to Evaluate the Safety and the Feasibility of Planning and Execution of Surgical Revascularization in Patients With Complex Coronary Artery Disease, Based Solely on MSCT Imaging Utilizing GE Healthcare Revolution CT and HeartFlow FFRCT.
Acronym: CABGRevolution
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Administrative issues
Sponsor: ECRI bv (Industry)
Collaborators: GE Healthcare (Industry); HeartFlow, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ECRI-12
Record Dates: First submitted 2019-02-12; First posted 2019-02-22 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Multivessel Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with 3-vessels diseased referred to CABG surgery (Other): Patients with 3-vessel disease (with or without left main involvement) for which the regular and conventional Heart Team has made already the decision to refer the patient for CABG treatment.
  Interventions: Radiation: Multi-sliced computed tomography (MSCT)

INTERVENTIONS:
Radiation: Multi-sliced computed tomography (MSCT) — Surgery planning done based solely on MSCT.

SUMMARY:
The CABG-REVOLUTION study is an investigator-initiated single-arm, multicentre, prospective study for patients with 3-vessel disease (with or without left-main involvement) referred to CABG treatment. Surgical revascularization strategy and treatment planning will be solely based on MSCT (with FFRCT) without knowledge of the anatomy defined by conventional cine-angiography.

DETAILED DESCRIPTION:
The CABG-REVOLUTION study is an investigator-initiated single-arm, multicentre, prospective study for patients with 3-vessel disease (with or without left-main involvement) referred to CABG treatment. Surgical revascularization strategy and treatment planning will be solely based on MSCT (with FFRCT) without knowledge of the anatomy defined by conventional cine-angiography.

One clinical follow-up visit including MSCT acquisition will be performed at 30 days after bypass surgery in order to assess graft patency and adequacy of the revascularization with respect to the surgical planning based on non-invasive imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Patient referred to CABG treatment (as assessed by 'conventional Heart Team');
2. Patients with at least 1 stenosis (visually determined de novo lesions with ≥50% DS) in all 3 major epicardial territories (LAD and/or side branch, CX and/or side branch, RCA and/or side branch) supplying viable myocardium with or without left main involvement;
3. Patients with hypoplastic right coronary artery (RCA) with absence of descending posterior and presence of a lesion in the LAD and circumflex (CX)territories may be included in the trial as a 3vessel disease equivalent. Ostial LAD plus ostial left circumflex artery (LCX) may be included in the trial as a Left Main equivalent
4. Distal vessel size should be at least 1.5 mm in diameter as visually assessed in diagnostic angiogram;
5. Patient with silent ischemia, chronic stable angina or stabilized acute coronary syndromes with normalized (stable or decreasing) cardiac biomarker values Note: For patients showing elevated Troponin (cTn) (e.g. non-STEMI patients) at baseline (within 24h pre-CABG) an additional blood sample must be collected prior to the CABG procedure to confirm that: • hs-cTn or Troponin I or T levels are stable, i.e. the value should be within 20% range of the value found in the first sample at baseline, or have dropped • CK-MB and CK levels are within normal range If hs-cTn or Troponin I or T levels are stable or have dropped, or the Creatine kinase-MB (CK-MB) and Creatine kinase (CK) levels are within normal ranges, and the ECG is normal, the patient may be included in the study.
6. All anatomical SYNTAX Scores are eligible;
7. Patient amenable to a MSCT coronary angiography (e.g. no claustrophobia, high heartrate not amenable to beta-blockers, poor renal function, etc., up to discretion of investigator);
8. Patient has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as approved by the Ethical Committee of the respective clinical site;
9. The patient agrees to the 1-month follow-up visit including a MSCT coronary angiography.

Exclusion Criteria:

1. Under the age of 18 years;
2. Unable to give Informed Consent;
3. Known pregnancy at time of enrollment. Female of childbearing potential i.e. who are not surgically sterile or post-menopausal (defined as no menses for 2 years without an alternative cause). Female who is breastfeeding at time of enrollment;
4. Prior percutaneous coronary intervention (PCI) or CABG; history of coronary stent implantation;
5. Evidence of evolving or ongoing acute myocardial infarction (AMI) in ECG and/or elevated cardiac biomarkers (according to local standard hospital practice);
6. Known renal insufficiency (e.g. serum creatinine >2.5mg/dL, or creatinine clearance ≤30 mL/min), or subject on dialysis, or acute kidney failure (as per physician judgment);
7. Concomitant cardiac valve disease requiring surgical therapy (reconstruction or replacement) and/or aneurysmectomy;
8. Single or two-vessel disease (at time of the conventional Heart Team consensus);
9. Non-graftable distal bed in >1 vessel as assessed by the surgeon based on conventional angiography;
10. Atrial fibrillation or significant arrhythmias;
11. Known allergy to iodinated contrast;
12. A Body Mass Index (BMI) of 35 or greater;
13. Currently participating in another trial and not yet at its primary endpoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2020-03-30 (Estimated); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients in the intention to treat (ITT) population for whom CABG planning and execution was based solely on MSCT. | 2 weeks after enrollment
Number of graft/anastomoses for which graft/anastomosis stenosis (≥50%DS - 99%DS) or occlusion (100%DS) occurred as percentage of the total number of intra graft/anastomoses. | 1 month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Patrick W Serruys, Prof. dr., Study Chair — NHLI Imperial College, London
Locations (4):
- University Hospital of Brussels, Brussels, Belgium
- University Hospital of Jena, Jena, Germany
- Centro Cardiologico Monzino, Milan, Italy
- University Hospital of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
The research data will be entered on separate forms and stored under a code number, according to prevailing legal requirements. No names or other personal data will be stored. Only the study doctor will hold the information to link the code to the patients. The encoded data will be processed, analysed and reported by the research employees of this study, who have an obligation of secrecy.
  Representatives of the sponsor or members of the Ethics Committee (EC) and regulatory authorities within Europe can have access to the medical files in order to inspect the correctness of the research data. Data may be provided to representatives and affiliates of the industries supporting the study: General Electric and HeartFlow Inc. It is possible that the results of this study are presented or published in medical journals; this will always be without mention of the identity of the patients.